CLINICAL TRIAL: NCT03292263
Title: Autologous Stem Cell Transplantation With Nivolumab in Patients With Multiple Myeloma
Brief Title: ASCT With Nivolumab in Patients With Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, R.M.Gorbacheva memorial institute vice director for research, St. Petersburg State Pavlov Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11/17-n
Record Dates: First submitted 2017-09-21; First posted 2017-09-25 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Nivolumab; Melphalan; Autologous hematopoietic stem cell transplantation
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mel+Nivo (Experimental): Autologous Stem Cell Transplant Drug: Melphalan 140-200 mg/m^2, Nivolumab100 mg iv days -3, +17
  Interventions: Drug: Melphalan; Drug: Nivolumab; Procedure: Autologous Stem Cell Transplantation

INTERVENTIONS:
Drug: Melphalan — iv infusion 70-100 mg/m2 on day -3, -2
  Other Names: Alkeran
Drug: Nivolumab — iv infusion 100 mg on day -3, +17
  Other Names: Opdivo
Procedure: Autologous Stem Cell Transplantation — peripheral blood stem cell transfusion at day 0

SUMMARY:
This is an open-label, single center trial of Autologous Stem Cell Transplantation (ASCT) with nivolumab in multiple myeloma patients to determine the efficacy and safety of ASCT and PD1 inhibitor combination.

For this purpose, 30 multiple myeloma patients, who have received induction therapy and have achieved a partial response (PR), stable disease (SD) or progression, and thus have unfavorable prognosis, will be treated with nivolumab administered iv at a dose of 100 mg on days 3 before and 17 after high-dose melphalan with autologous stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with MM (Multiple Myeloma)
* Partial response, stable disease or progression after induction therapy (including ASCT)
* Measurable disease
* Successful peripheral blood stem cell collection with G-CSF
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2
* Signed informed consent
* Patients after first-line induction therapy

Exclusion Criteria:

* Another malignancy requiring treatment at the time of inclusion
* History of interstitial lung disease or pneumonitis
* Patients with any other known concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes; cardiovascular disease including congestive heart failure NYHA Class III or IV, myocardial infarction within 6 months, and poorly controlled hypertension) which, in the opinion of the investigator could compromise participation in the study
* Uncontrolled bacterial or fungal infection at the time of enrollment
* Pregnancy
* Somatic or psychiatric disorder making the patient unable to sign informed consent
* Active or prior documented autoimmune disease requiring systemic treatment
* Prior treatment with anti-PD-1, anti-PD-L1, or anti-CTLA4 therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-04-24 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall response | 3 months
  Includes complete response, very good partial response, and partial response (based on IMWG criteria)

SECONDARY OUTCOMES:
Progression free survival (PFS) | 12 months
  PFS will be assessed with Kaplan-Meier method from the date of ASCT, with day 0 defined as date of stem cell infusion (in case of tandem transplant the 2nd of 2 transplants will be used) until the date of progression, defined as the date at which the patient starts the next line of therapy or the date of death.
Overall Survival (OS) | 24 months
  Will be assessed with Kaplan-Meier method from the date of ASCT, with day 0 defined as date of stem cell infusion (in case of tandem transplant the 2nd of 2 transplants will be used)
Frequency of grade 3 or higher treatment-related adverse events by CTCAE 4.03 | 12 months
  Toxicity parameters based on NCI CTCAE 4.03 grades: hematological toxicity (CBC), hepatotoxicity (liver function tests), nephrotoxicity (creatinine), neurotoxicity (attending physician assessment), fatigue (attending physician assessment), rash (attending physician assessment), colitis (attending physician assessment), pneumonitis (attending physician assessment), autoimmune disorders (level of hormones, presence of autoimmune antibodies, attending physician assessment).

CONTACTS AND LOCATIONS:
Locations (1):
- Boris V Afanasyev, MD, Prof., Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided